CLINICAL TRIAL: NCT02731846
Title: A Phase III, 4-week, Randomized, Double-blind Study to Compare 'Closed' Triple Therapy (FF/UMEC/VI), 'Open' Triple Therapy (FF/VI + UMEC) and Dual Therapy (FF/VI) in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study Comparing the Closed Triple Therapy, Open Triple Therapy and a Dual Therapy for Effect on Lung Function in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: It has been determined on June 10th that the 205165 study will not progress. This decision has been made prior to study start, no patients were screened.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205165
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Efficacy; Triple therapy; Parallel; Respiratory
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; GSK573719; vilanterol; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FF/UMEC/VI (100/62.5/25 mcg) + placebo (Experimental): Subjects will receive FF/UMEC/VI 100 mcg/62.5 mcg/25 mcg delivered via single ELLIPTA inhaler ('closed' triple) and matching placebo via ELLIPTA inhaler once daily in the morning for 4 weeks as per the randomization. Albuterol/salbutamol will be used as rescue medication throughout the study as needed.
  Interventions: Drug: Fluticasone furoate 100 mcg + Umeclidinium 62.5 mcg+Vilanterol 25 mcg; Drug: Fluticasone furoate 100 mcg + Vilanterol 25 mcg; Drug: Umeclidinium 62.5 mcg; Device: Placebo ELLIPTA inhaler; Drug: Albuterol/Salbutamol
- FF/VI 100 mcg/25 mcg + UMEC 62.5 mcg (Experimental): Subjects will receive FF/VI (100 mcg/25 mcg) and UMEC 62.5 mcg delivered via two ELLIPTA inhaler ('open' triple) once daily in the morning for 4 weeks as per the randomization. Albuterol/salbutamol will be used as rescue medication throughout the study as needed.
  Interventions: Drug: Fluticasone furoate 100 mcg + Umeclidinium 62.5 mcg+Vilanterol 25 mcg; Drug: Fluticasone furoate 100 mcg + Vilanterol 25 mcg; Drug: Umeclidinium 62.5 mcg; Drug: Albuterol/Salbutamol
- FF/VI 100 mcg/25 mcg + placebo (Experimental): Subjects will receive FF/ VI (100 mcg/25 mcg) delivered via single ELLIPTA inhaler and matching placebo via ELLIPTA inhaler once daily in the morning for 4 weeks as per the randomization. Albuterol/salbutamol will be used as rescue medication throughout the study as needed.
  Interventions: Drug: Fluticasone furoate 100 mcg + Vilanterol 25 mcg; Device: Placebo ELLIPTA inhaler; Drug: Albuterol/Salbutamol

INTERVENTIONS:
Drug: Fluticasone furoate 100 mcg + Umeclidinium 62.5 mcg+Vilanterol 25 mcg — Dry white powder delivered via ELLIPTA inhaler(2 strips with 30 blisters each, first containing fluticasone furoate 100 mcg per blister and second containing Umeclidinium 62.5 mcg and Vilanterol 25 mcg per blister), administered as one inhalation of FF/UMEC/VI (100/62.5/25 mcg) once-daily in the morning
  Arms: FF/UMEC/VI (100/62.5/25 mcg) + placebo; FF/VI 100 mcg/25 mcg + UMEC 62.5 mcg
Drug: Fluticasone furoate 100 mcg + Vilanterol 25 mcg — Dry white powder delivered via ELLIPTA inhaler (2 strips with 30 blisters each, first containing fluticasone furoate 100 mcg per blister and second containing Vilanterol 25 mcg per blister), administered as one inhalation of FF/VI (100/25 mcg) once-daily in the morning
Drug: Umeclidinium 62.5 mcg — Dry white powder delivered via ELLIPTA inhaler (1 strip with 30 blisters containing Umeclidinium 62.5 mcg, administered as one inhalation once-daily in the morning
  Arms: FF/UMEC/VI (100/62.5/25 mcg) + placebo; FF/VI 100 mcg/25 mcg + UMEC 62.5 mcg
Device: Placebo ELLIPTA inhaler — Placebo will be administered via ELLIPTA inhaler. Dry white powder administered as one inhalation each morning (1 strip with 30 blisters containing placebo)
  Arms: FF/UMEC/VI (100/62.5/25 mcg) + placebo; FF/VI 100 mcg/25 mcg + placebo
Drug: Albuterol/Salbutamol — Albuterol/salbutamol will be administered via metered-dose inhaler (MDI) with a spacer as needed throughout the study as a rescue medication

SUMMARY:
The primary purpose of this study is to assess the equivalence of closed triple therapy Fluticasone Furoate (FF)/Umeclidinium (UMEC)/Vilanterol (VI) to open triple therapy (FF/VI + UMEC), with a comparison of both triple therapies to dual therapy (FF/VI) on lung function.

This is a phase III, 4-week, randomized, double-blind, parallel group, multicenter study comparing FF/UMEC/VI (100 micrograms [mcg]/62.5 mcg/25 mcg) delivered via a single ELLIPTA® inhaler ('closed' triple) + matching placebo ELLIPTA inhaler, FF/VI + UMEC delivered via two ELLIPTA inhalers ('open' triple) and FF/VI via a single ELLIPTA inhaler + matching placebo ELLIPTA inhaler, all once daily. The total duration of subject participation will be approximately 7 weeks, consisting of a 2-week run-in period, 4-week treatment period and a 1-week follow-up period.

ELLIPTA is a registered trade mark of the GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated written informed consent prior to study participation.
* Outpatient
* Subjects 40 years of age or older at Screening (V1).
* Male or female subjects.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

  * Non-reproductive potential as defined in the protocol
  * Reproductive potential and agrees to follow methods specified in the protocol for avoiding pregnancy in Females of Reproductive Potential (FRP), from 30 days prior to the first dose of study treatment and until after the last dose of study treatment and completion of the follow-up visit.
* An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society
* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at Screening [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Screening (V1).
* A score of >=10 on the COPD Assessment Test (CAT) at Screening (V1).
* A post-albuterol/salbutamol FEV1/ forced vital capacity (FVC) ratio of <0.70 and a post-albuterol/salbutamol FEV1 of =<70 percent of predicted normal values at Screening (V1).

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD, which is the primary cause of their respiratory symptoms).
* Subjects with alpha-1-antitrypsin deficiency as the underlying cause of COPD.
* Subjects with active tuberculosis are excluded. Subjects with other respiratory disorders (e.g. clinically significant: bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases) are excluded if these conditions are the primary cause of their respiratory symptoms.
* Subjects with lung volume reduction surgery (including procedures such as endobronchial valves) within the 12 months prior to Screening (V1).
* Immune suppression (e.g. advanced Human Immunodeficiency Virus (HIV) with high viral load and low CD4 count, Lupus on immunosuppressants that would increase risk of pneumonia) or other risk factors for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis).subjects at potentially high risk for pneumonia (e.g. very low BMI, severely malnourished, or very low FEV1) will only be included at the discretion of the investigator.
* Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening (V1) and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable).
* Other respiratory tract infections that have not resolved at least 7 days prior to Screening (V1).
* Chest x-ray reveals evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD, or another condition that would hinder the ability to detect an infiltrate on chest x-ray (e.g. significant cardiomegaly, pleural effusion or scarring). All subjects will have a chest x-ray at Screening (V1) [or historical radiograph or CT scan obtained within 12 months prior to Screening. Subjects who have experienced pneumonia and/or moderate or severe COPD exacerbation within 12 months of Screening (V1) must provide a post pneumonia/exacerbation chest x-ray or have a chest x-ray conducted at Screening (V1)].

  • For sites in Germany: If a chest x-ray (or CT scan) within 12 months prior to Screening (V1) is not available, approval to conduct a diagnostic chest x-ray will need to be obtained from the Federal Office for Radiation Protection (BfS).
* Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Alanine aminotransferase (ALT) >2x upper limit of normal (ULN); and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* Subjects with any of the following at Screening (V1) are excluded:

  * Myocardial infarction or unstable angina in the last 6 months
  * Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months
  * New York Heart Association Class IV Heart failure
* Abnormal and clinically significant 12-Lead electrocardiogram (ECG) finding. An abnormal and clinically significant finding that would preclude a subject from entering the trial is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following:

  * Atrial fibrillation with rapid ventricular rate >120 beats per minute;
  * Sustained or non sustained ventricular tachycardia;
  * Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted).
* A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the investigator, contraindicates study participation.
* Subjects with carcinoma that has not been in complete remission for at least 3 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 3 year waiting period if the subject has been considered cured by treatment.
* Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3 liter (L)/min (Oxygen use =<3 L/min flow is not exclusionary)
* Subjects who are medically unable to withhold their albuterol/salbutamol for the 4-hour period required prior to spirometry testing at each study visit.
* Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete study related materials.
* Use of the below medications within the specified time intervals prior to Screening (V1): 1.Long term continuous antibiotic therapy for >= 30 days 2.Systemic, Oral, parenteral corticosteroids 3.Any other investigational drug

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in trough forced expiratory volume in one second (FEV1) on Day 29 | Up to Day 29
  Forced Expiratory Volume (FEV1) is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second

SECONDARY OUTCOMES:
Change from baseline in trough FEV1 on Day 2 and Day 28 | Up to Day 28
  Change from baseline in trough FEV1 will be evaluated to compare the effect of FF/UMEC/VI with FF/VI + UMEC
Change from baseline in trough FEV1 on Days 2, 28 and 29 | Up to Day 29
  Change from baseline in trough FEV1 will be evaluated to compare the effect of FF/UMEC/VI and FF/VI + UMEC with FF/VI
Change from baseline in weighted mean (WM) FEV1 0-6 hours on Day 1 and Day 28 (in a subset) | Up to Day 28
  Change from baseline in weighted mean FEV1 0-6 hours will be evaluated to compare the effect of FF/UMEC/VI with FF/VI + UMEC and also to compare the effect of FF/UMEC/VI and FF/VI + UMEC with FF/VI
Serial FEV1 over 0-6 hours on Day 1 and Day 28 (in a subset) | Up to Day 28
  Serial FEV1 over 0-6 hours will be evaluated to compare the effect of FF/UMEC/VI with FF/VI + UMEC and also to compare the effect of FF/UMEC/VI and FF/VI + UMEC with FF/VI

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Canada (3):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- Germany (2):
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin